CLINICAL TRIAL: NCT02212184
Title: Diaphragm Release Manual Technique Efficacy on Diaphragmatic Mobility, Respiratory Muscle Strength and Exercise Performance in COPD Patients: a Randomized Controlled Trial
Brief Title: Diaphragm Release Manual Technique Efficacy in COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helga Cecília Muniz de Souza (Other)
Collaborators: Universidade Federal de Pernambuco (Other)
Responsible Party: Sponsor-Investigator, Helga Cecília Muniz de Souza, MsC, Universidade Federal de Pernambuco
Organization: Universidade Federal de Pernambuco (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Manual Therapy in COPD
Record Dates: First submitted 2014-06-12; First posted 2014-08-08 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: COPD
Keywords: Diaphragm; COPD; Musculoskeletal Manipulations; Ultrasonography; Optoelectronic Plethysmography.
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Sham Comparator): Manual Diaphragm release technique (sham) In attempt to execute the sham protocol the therapist performs manual contact (pisiform, ulnar edge and the last three fingers) with the underside of the costal cartilage of the 7th, 8th, 9th and 10th rib. The therapist will hold only light touch in the landmarks, without exerting pressure or traction. The maneuver will be performed in two sets of ten deep breaths, with an one minute interval between them.
  Interventions: Other: Manual Diaphragm release technique (sham)
- Intevention Group (Experimental): All patients will receive the Manual Diaphragm Release Technique, during 6 days of treatment. They will undertake four evaluations throughout treatment: before and immediately after the Day 1 (Baseline 1 and Post 1) and before and after Day 6 (Baseline 6 and Post 6).
  In the other Days (2nd to 5th) patients will only receive the intervention and won't be evaluated.
  Interventions: Other: Manual Diaphragm Release Technique

INTERVENTIONS:
Other: Manual Diaphragm Release Technique — The therapist performs manual contact (pisiform, ulnar edge and the last three fingers) with the underside of the costal cartilage of the 7th, 8th, 9th and 10th rib, and guiding forearms toward the shoulders of the corresponding side. During inspiration, pulls the points of contact with both hands, in the direction of the head, accompanying the elevation movement of the ribs. During exhalation, deepens contact toward the inner costal, maintaining resistance. 2 sets x 10 breaths (1 min interval). Treatment will last two weeks (6 sessions) All patients will undertake four evaluations throughout treatment: Baseline Day 1 and post Day 1; Baseline Day 6 and post Day 6.
  Other Names: Manual Diaphragm Stretching Technique
  Arms: Intevention Group
Other: Manual Diaphragm release technique (sham) — Manual Diaphragm release technique (sham) In attempt to execute the sham protocol the therapist performs manual contact (pisiform, ulnar edge and the last three fingers) with the underside of the costal cartilage of the 7th, 8th, 9th and 10th rib. The therapist will hold only light touch in the landmarks, without exerting pressure or traction. The maneuver will be performed in two sets of ten deep breaths, with an one minute interval between them.
  Arms: Control Group

SUMMARY:
The aims of this study are to evaluate the effects of Diaphragm Release Manual Technique on diaphragm mobility, chest wall kinematics and functional capacity of COPD patients. Methods: Randomized controlled trial (double blinded) with COPD patients, allocated in two group: intervention (IG) who will receive the Diaphragm Release manual technique on 6 non-consecutive sessions and control group (CG), who will receive a sham protocol (light touch) with the same parameters of IG. Outcomes will be evaluated as: immediate and post treatment effects (after 1 and 6 sessions respectively). The primary outcome analysed will be the diaphragm displacement (ultrasonography evaluation) and secondary outcomes will comprise abdominal and chest wall kinematics.

ELIGIBILITY:
Inclusion Criteria:

* CPOD patients
* ex-smokers
* clinically stable patients (no exacerbation in the previous 6 weeks)
* forced expiratory volume in one second (FEV1) < than 80% predicted
* FEV1/FVC ≤ 0.7, post bronchodilator

Exclusion Criteria:

* cardiopulmonary diseases
* BMI > 30.0 kg/m2
* History of thoracic surgery
* Denial to participate

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Diaphragm mobility | Diaphragm mobility at first session and after two weeks of treatment.
  To evaluate diaphragmatic mobility a high-resolution ultrasound SonoaceR3 (Samsung Medison - South Korea) with a 3.5 MHz convex transducer will be used. Volunteers will remain in a supine position and receive verbal command to perform Inspiratory capacity maneuvers (IC), and the measurement of each curve referring to the diaphragmatic displacement (in mm) will be performed immediately after obtaining the images. The maneuvers will be repeated until obtaining 5 satisfactory images. The average of the three highest values not differing by more than 10% between their values should be accepted.

SECONDARY OUTCOMES:
Compartmental Chest wall volume | Compartmental Chest wall volume evaluated by Opto-electronic Plethysmograph at the first session and after two weeks of treatment
  Compartmental Chest wall volume will be measured by Opto-electronic Plethysmograph (OEP) (BTS Bioengineering, Italy) with 89 reflective markers placed on volunteer´s skin surface using a hypoallergenic adhesive on specific anatomical points of the chest wall and abdomen. Thus, changes in chest wall volumes are going to be calculated, allowing to acquire total chest wall volume (Vcw) and the division into three compartments, namely: pulmonary rib cage (Rc,p), abdominal rib cage (Rc,a) and abdomen (Ab) during quiet breathing, inspiratory capacity (IC) and vital capacity (VC), maneuvers.

OTHER OUTCOMES:
Six-minute walking distance | Six-minute walking distance (6MWD) evaluated by 6 minutes walking test at the first session and after two weeks of treatment
  Six-minute walking tests (6MWT) will be performed in accordance to the ATS/ERS criteria, in the moments: Pre 1st session and Pre 6th session.
Respiratory muscle strength | Respiratory muscle strength measured by manovacuometry at the first session and after two weeks of treatment
  Maximum inspiratory and expiratory pressures (MIP, MEP) will be obtained from the residual volume and total lung capacity, respectively, according to ATS/ERS criteria using a portable digital manometer, model MVD 300 (® MDI Ltda, Brazil). With the same instrument, the patient's nasal inspiratory pressure (SNIP) will also be assessed by placing the nasal plug into one nostril, without contralateral occlusion. Ten Sniff maneuvers should be performed with maximal inspiratory effort (60 seconds between each) and the greatest value achieved will be considered.

CONTACTS AND LOCATIONS:
Overall Officials: Armele D de Andrade, Post Doctor, Study Director — Universidade Federal de Pernambuco
Locations (1):
- UFPernambuco, Recife, Pernambuco, Brazil

REFERENCES:
- [Derived] Rocha T, Souza H, Brandao DC, Rattes C, Ribeiro L, Campos SL, Aliverti A, de Andrade AD. The Manual Diaphragm Release Technique improves diaphragmatic mobility, inspiratory capacity and exercise capacity in people with chronic obstructive pulmonary disease: a randomised trial. J Physiother. 2015 Oct;61(4):182-9. doi: 10.1016/j.jphys.2015.08.009. Epub 2015 Sep 19. PMID 26386894